CLINICAL TRIAL: NCT05807854
Title: Treatment of Degenerative Massive Rotator Cuff Tears: a Multicenter, Randomized Comparative Surgical Trial
Brief Title: RSA Vs RCR for Massive RCTs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: La Tour Hospital (Other)
Responsible Party: Principal Investigator, Dr. Alexandre Lädermann, Orthopaedic Surgeon FMH, Shoulder and Elbow Surgery Traumatology, La Tour Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-00111
Record Dates: First submitted 2023-03-29; First posted 2023-04-11 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Rotator Cuff Tears
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Arthroscopy

STUDY DESIGN:
Intervention Model Description: Multicenter, Randomized Comparative Surgical Trial
Masking Description: The statistician will be blinded to patient allocation groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Arthroscopic surgery (Active Comparator): The massive degenerative rotator cuff tear are treated by arthroscopy. It consists in reattaching the torn tendon with anchors and sutures.
  Interventions: Procedure: Arthroscopy
- Reverse shoulder arthroplasty (Experimental): The problems induced by the massive degenerative rotator cuff tear are solved by a complete replacement of the shoulder joint with a prosthesis (reverse design).
  Interventions: Device: Reverse Shoulder Arthroplasty

INTERVENTIONS:
Procedure: Arthroscopy — The surgeon reattaches the torn tendon to the bone with anchors and sutures.
  Arms: Arthroscopic surgery
Device: Reverse Shoulder Arthroplasty — It consists in replacing the shoulder joint with a total shoulder prosthesis (reverse design).
  Arms: Reverse shoulder arthroplasty

SUMMARY:
Different treatment options are available for massive or irreparable rotator cuff tears. An arthroscopic or an open repair approach is possible in the majority of cases and functional outcomes are improved, particularly when a complete arthroscopic repair can be achieved. However, the healing rate of massive rotator cuff tears after repair may remain low and failure of healing is associated with progression of arthritis. An alternative to arthroscopic or open repair is reverse shoulder arthroplasty which decreases pain and improves function, active shoulder elevation and quality of life. The primary goal of this prospective multicentric randomized study is to determine if there is a difference of functional outcomes between rotator cuff repair (RCR) repair and reverse shoulder arthroplasty (RSA).

DETAILED DESCRIPTION:
The majority of degenerative rotator cuff tears occur in individuals over 60 years of age. Therefore, as our population increases in size and advances in age, the incidence of rotator cuff tears is also increasing. A growing number of people are remaining active at this age, and continue to place substantial physical demands on their shoulders notably into their seventh and eighth decades of life. At the same time, the rotator cuff undergoes intrinsic degeneration and the prevalence of osteoporosis increases. Consequently, a significant and growing number of arthroscopic rotator cuff repairs are performed in individuals with poor soft tissue or bone quality. Moreover, whereas most rotator cuff tears occur at the tendon-bone insertion, fixation quality can be challenged by a tear that occurs more medially, leaving only a small amount of tendon for fixation by suture.

Different treatment options are available for massive or irreparable rotator cuff tears, including debridement and subacromial decompression, repair (partial or complete), transfer of the subscapularis tendon, transfer of the teres major muscle, deltoid flap reconstruction, transfer of the latissimus dorsi or the pectoralis major, superior capsule reconstruction, augmented cuff repair, subacromial balloon and reverse total shoulder replacements. None of these treatments has proved superiority on other ones, particularly when the rotator cuff is massively torn.

Massive degenerative rotator ruff tears are a challenge. An arthroscopic or an open repair approach is possible in the majority of cases and functional outcomes are improved, particularly when a complete arthroscopic repair can be achieved. However, the healing rate of massive rotator cuff tears after repair may remain low and failure of healing is associated with progression of arthritis. An alternative to arthroscopic or open repair is reverse shoulder arthroplasty which decreases pain and improves function, active shoulder elevation and quality of life. Recently, Liu et al. demonstrated that both rotator cuff repair (RCR) and reverse shoulder arthroplasty (RSA) are effective and reliable options for massive rotator cuff tears (RCT), but revealed a better shoulder function for patients in the rotator cuff repair (RCR) group. While these results are interesting, this study remains retrospective and call for new studies with a higher level of evidence.

The primary goal of this prospective multicentric randomized study is to determine if there is a difference of functional outcomes between rotator cuff repair (RCR) repair and reverse shoulder arthroplasty (RSA).

ELIGIBILITY:
Inclusion Criteria:

* 1 Patient voluntarily consents to participate
* 2 Patient with a massive and reparable non traumatic rotator cuff tears after failure of conservative treatment
* 3 Patients with the following pre-operative images: Three standardized X-rays series and Magnetic Resonance Imaging (MRI) or arthro Magnetic Resonance Imaging without sign of traumatic lesions

Exclusion Criteria:

* 1 Patient has known intentions, obligations, or co-morbidity that would inhibit them from participating in the study
* 2 Revision rotator cuff repair
* 3 Patient consent withdrawal
* 4 Glenohumeral arthritis defined as stage > 3 Hamada classification
* 5 Infection and neuropathic joints
* 6 Known or suspected non-compliance, drug or alcohol abuse
* 7 Patients incapable of judgement or under tutelage
* 8 Inability to follow the procedures of the study
* 9 Enrolment of the investigator, his/her family members, employees and other dependent persons

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
American Shoulder and Elbow Surgeon (ASES) score | At 24 post-operative months
  American Shoulder and Elbow Surgeon (ASES) score. From 0 (worst) to 100 (best).

SECONDARY OUTCOMES:
Pain on Visual Analogue Scale (pVAS) | At 24 post-operative months
  Pain on Visual Analogue Scale (pVAS). From 0 (best) to 10 (worst)
Constant score | At 24 post-operative months
  From 0 (worst) to 100 (best)
Single Assessment Numeric Evaluation (SANE) | At 24 post-operative months
  Single Assessment Numeric Evaluation (SANE). From 0 (worst) to best (100)
Complication | Within the 24 post-operative months
  Any type of post-operative or intra-operative complication
Location of the defect | At 24 post-operative months
  (at the foot print | medial cuff failure). Radiographic outcome evaluated using an ultrasound examination. Only for the Arthroscopic group.
Signs of anchor displacement and location | At 24 post-operative months
  (lateral | medial row). Radiographic outcome evaluated using an ultrasound examination. Only for the Arthroscopic group.
Signs of suture cut-through | At 24 post-operative months
  (yes | no). Radiographic outcome evaluated using an ultrasound examination. Only for the Arthroscopic group.
Patient satisfaction | At 24 post-operative months
  Licker scale comprising 7 points
Range of motion | At 24 post-operative months
  Passive and active
Tendon defect | At 24 post-operative months
  According to the Sugaya classification
Signs of stem or glenoid loosening | At 24 post-operative months
  X-ray evaluation
Scapular notching | At 24 post-operative months
  X-ray evaluation
Dislocation | At 24 post-operative months
  X-ray evaluation
Acromial fracture | At 24 post-operative months
  X-ray evaluation
Stem subsidence | At 24 post-operative months
  X-ray evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Lädermann, MD, Principal Investigator — La Tour hospital, Meyrin (1217) Geneva, Switzerland; Patrick Denard, MD, Principal Investigator — Department of Orthopaedics and Rehabilitation, Oregon Health & Science University, Portland, OR, USA
Locations (2):
- Oregon Health & Science University, Portland, Oregon, United States
- La Tour hospital, Meyrin, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
Under reasonable request from scientists (with accepted research protocol)

REFERENCES:
- [Derived] Ladermann A, Pernoud A, Cochard B, Bothorel H. Treatment of degenerative massive rotator cuff tears: a study protocol for a randomized non-inferiority comparative surgical trial. Trials. 2025 Aug 4;26(1):270. doi: 10.1186/s13063-025-08990-9. PMID 40759980